CLINICAL TRIAL: NCT07151508
Title: Successful Treatment of Netherton Syndrome With Combination of Secukinumab and Dupilumab.
Status: Completed | Type: Observational
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCHPOI-2025--07
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Neterton Syndrome
Keywords: Neterton syndrome; targeted treatment; secukinumab; dupilumab; ichtiosis; atopy; IL-17; IL-4/13

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Secukinumab was administered in a weight-adapted dosing regimen ? Dupilumab was administered at a dose dependent on the patient's weight and age — Secukinumab was administered in a weight-adapted dosing regimen equivalent to that used in clinical trials for psoriasis: 75 mg for less than 25 kg,150 mg for 25 to 50 kg, and 300 mg for greater than 50 kg at baseline and weeks1,2,3, and 4 and monthly there after.
  Dupilumab was administered at a dose dependent on the patient's weight and age in accordance with the instructions.

SUMMARY:
In this study, we describe our experience with secukinumab (IL-17A inhibitor) and dupilumab (IL-4/IL-13 inhibitor) treatment of a group of pediatric patients with severe Neterton syndrome.

DETAILED DESCRIPTION:
Pediatric patients qualified for participation in the study if they had a documented diagnosis of Neterton syndrome and they received treatment with sekukinumab or dupilumab for at least 3 months.

All patients received treatment in the Department of Immunology at the Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology from January 2021 to June 2024.

A total of 15 patients from 13 families with NS were enrolled in the study. The median age of the patients was 8 years (1;15), and the male/female ratio 9/6.

In this study, 14 patients initially received secukinumab therapy, for 12/14 patients dupilumab was added, and 2 patients continued secukinumab monotherapy. The median time to switch from secukinumab monotherapy to combination therapy was 4 months (3;27). One patient initially received dupilumab monotherapy and was switched to combination therapy (Fig. 1). Treatment duration for each type of treatment was at least 3 months at the time of this report.

Secukinumab was administered in a weight-adapted dosing regimen equivalent to that used in clinical trials for psoriasis: 75 mg for less than 25 kg,150 mg for 25 to 50 kg, and 300 mg for greater than 50 kg at baseline and weeks1,2,3, and 4 and monthly there after.

Dupilumab was administered at a dose dependent on the patient's weight and age in accordance with the instructions.

The patients were evaluated before and 3-6 months after treatment initiation of secukinumab/dupilumab and combination therapy, including laboratory monitoring of complete blood cell count, liver enzyme levels, kidney function tests and IL17A levels in CD4 lymphocytes. Treatment response was assessed by the following criteria: ISS total score, IgE level and and IL17A levels in CD4 lymphocytes.

Additionally, standardized photographs were taken by a medical photographer. The ISS total score was assessed on these photographs.

All adverse events (AEs) during therapy were recorded. The investigator provided guidance to the patient or caregiver on how to identify and document AEs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with Neterton syndrome
* Treatment with secukinumab and/or dupilumab for at least 3 months

Exclusion Criteria:

* Irregular administration of therapy
* Development of a serious adverse event

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with Neterton syndrome
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
overal survival Kaplan-Mayer method | 3 and 6 months from the start of each type of therapy
  Evaluation of the efficacy and safety of dupilumab and secukinumab therapy in patients with Netherton syndrome

SECONDARY OUTCOMES:
event free survival | 3 and 6 months from the start of each type of therapy
  Evaluation of the efficacy and safety of dupilumab and secukinumab therapy in patients with Netherton syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, Russia